CLINICAL TRIAL: NCT02120495
Title: Application of Digital Techniques in Intraoral Condylectomy Via Coronoid Process Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, wang xiaoxia, associate professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: wxiaoxia1
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Surgical Approach & Incisions
Keywords: condylectomy; TMJ function; intraoral approach
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intraoral condylectomy via coronoid process resction (Experimental): This procedure has no facial nerve injury and skin scar,little injury to TMJ anatomy and function.
  Interventions: Procedure: condylectomy

INTERVENTIONS:
Procedure: condylectomy — The condylectomy via intraoral approach will avoid the risk of facial nerve injury and skin scar compared with the preauricular incision.And it can also greatly reserve the temporomandibular jiont anatomy and function.
  Other Names: surgical approach

SUMMARY:
This study will apply the digital techniques to do the condylectomy through an intraoral approach without needing to do the intraoral vertical ramus osteotomy (IVRO). This new surgical technique will greatly maintain the TMJ anatomy structure, reduce the risk and increase the precision of the operation procedure.

DETAILED DESCRIPTION:
In this study we will use the digital techniques such as pre-surgical visual treatment planning, real time surgical navigation system, endoscope techniques, to do the intraoral condylectomy via coronoid process resection. After the condyle lesion resection, the coronoid process will be reimplanted and fixed by stainless steel wire. By using these techniques we can safely and precisely cut proper size and position of the condyle lesion as we pre-surgically designed, and at the same time greatly maintain the temporomandibular joint anatomy structure. Since we don't need to do the mandible vertical ramus osteotomy, and no conventional extraoral incision will be needed, the surgical injury will be minimized and the TMJ function will recover soon postoperatively. Additionally, the intraoral approach can avoid the risk of facial nerve injury, salivary fistula and skin scar, so it has better aesthetic results than the preauricular approach and the submandibular approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandible condylar hyperplasia or osteoma who need to do the condylectomy to prevent the active growth of the affected mandible condyle and the consequence progressive facial asymmetry
* Usually the patients have TMJ functional disorder; and the SPECT shows difference greater than 20% (pixel count) between the affected side and the contralateral normal side.

Exclusion Criteria:

* Patients with contradictions to do the operation procedure and general anesthesia, patients refuse to accept the condylectomy, or patients can't afford the extra cost for the application of digital techniques are excluded from this study

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
complications of condylectomy | post-operative day 7 and 6 months
  to record the complications of the operation and the TMJ function recovering.

CONTACTS AND LOCATIONS:
Overall Officials: xiaoxia wang, MD, Principal Investigator — Peking University School of Stomatology
Locations (1):
- Peking University Hospital of Stomatology, South Zhongguancun Avenue22, Beijing Municipality, China